CLINICAL TRIAL: NCT05481788
Title: External Evaluation of Vancomycin Population Pharmacokinetic Models and Development of Continuous Infusion Dosing Recommendations
Brief Title: External Evaluation of Vancomycin Population Pharmacokinetic Models
Acronym: EOPMV
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: EOPMV - 29BRC21.0126
Record Dates: First submitted 2021-06-18; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Vancomycin Dosage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
All patients treated with vancomycin hospitalized outside of ICU in Brest University Hospital from 1rst january 2019 to 1rst january 2021 will be screened for inclusion. Vancomycin dosage, age, weight and serum creatinin will be recorded.

Seven pharmacokinetic models' predictive performance will be evaluated on this database.

Using the best model, we will perform Monte-Carlo simulation to elaborate dosing nomograms and develop dosing recommandations of continuous infusion of vancomycin.

DETAILED DESCRIPTION:
Monte Carlo simulations will be performed according to varying creatinin clearance values and weight, for both the loading dose and the maintenance dose.

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in Brest University Hospital,
* treated with vancomycin and receiving pharmacological monitoring
* between 1rst January 2019 and 1rst January 2021

Exclusion Criteria:

* Missing data on vancomycin administration
* Refusal to be included in this study
* Hospitalisation in ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults treated with vancomycin outside of ICU
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Imprecision in Predictive performance of seven pharmacokinetic models | September 2021
  The model with the lesser imprecision reported on the Observed vs Predicted Concentrations Graph will be selected
Bias in Predictive performance of seven pharmacokinetic models | September 2021
  The model with the lesser bias reported on the Observed vs Predicted Concentrations Graph will be selected

CONTACTS AND LOCATIONS:
Locations (1):
- Brest University Hospital, Brest, France